CLINICAL TRIAL: NCT03688074
Title: A Phase 2, Randomized, Double-blind, Parallel Group, Placebo Controlled Study to Evaluate the Effect of Tezepelumab on Airway Inflammation in Adults With Inadequately Controlled Asthma on Inhaled Corticosteroids and at Least One Additional Asthma Controller (CASCADE)
Brief Title: Study to Evaluate Tezepelumab on Airway Inflammation in Adults With Uncontrolled Asthma (CASCADE)
Acronym: CASCADE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5180C00013
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Results first posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Asthma; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases, Obstructive; Lung Diseases; Respiratory Hypersensitivity; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases
Keywords: Asthma; Uncontrolled asthma; Severe uncontrolled asthma
MeSH Terms: conditions — Asthma; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases, Obstructive; Lung Diseases; Respiratory Hypersensitivity; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases | interventions — tezepelumab

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 1:1 ratio to either tezepelumab or matching placebo both administered subcutaneously.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tezepelumab (Experimental): Tezepelumab subcutaneous injection
  Interventions: Biological: Tezepelumab
- Placebo (Placebo Comparator): Placebo subcutaneous injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Tezepelumab — Tezepelumab subcutaneous injection
  Arms: Tezepelumab
Other: Placebo — Placebo subcutaneous injection
  Arms: Placebo

SUMMARY:
A phase 2, multicentre, randomized, double-blind, placebo-controlled, parallel group study to evaluate the effect of tezepelumab on airway inflammation in adults with inadequately controlled asthma.

DETAILED DESCRIPTION:
This is a multicentre, randomized, double-blind, placebo-controlled, parallel group study to evaluate the effect of tezepelumab on airway inflammation in adults with inadequately controlled moderate-to-severe asthma, taking inhaled corticosteroids and at least one additional asthma controller. Approximately 110 subjects will be randomized globally. Subjects will receive tezepelumab, or placebo, administered via subcutaneous injection at the study site, over a 28-week treatment period. Although, due to the Covid-19 pandemic this may be an extended time frame for some subject visits. The study also includes a post-treatment follow-up period of 12 weeks.

ELIGIBILITY:
Principal Inclusion Criteria:

* Subject must be 18 to 75 years of age.
* Documented physician-diagnosed asthma for at least 12 months.
* Subjects who have received a physician- prescribed asthma controller medication with medium or high dose ICS for at least 12 months; must be stable for at least 3 months prior to screening visit.
* At least one additional maintenance asthma controller medication is required according to standard practice of care and must be documented for at least 3 months.
* At enrolment, the subject must have a predicted normal value for the morning pre-bronchodilator FEV1>50% and more than 1L.
* Evidence of asthma as documented by reversibility of FEV1 ≥12% and ≥200 mL in the previous 12 months prior to screening, or during the screening period prior to randomization.
* ACQ-6 score ≥ 1.5 during the screening period prior to randomization.

Principal Exclusion Criteria:

* Any clinically important pulmonary disease other than asthma.
* History of cancer.
* Hospitalization or required OCS for asthma exacerbation within 6 weeks of enrolment or >3 exacerbations requiring OCS or hospitalization in the year prior to visit 1 or who had been intubated or admitted to ICU for asthma exacerbation in the year prior to enrolment.
* History of a clinically significant infection, including upper (URTI) or lower respiratory tract infection (LRTI), requiring treatment with antibiotics or antiviral medications finalized <2 weeks before visit 1 or during the run-in period.
* Current smokers or subjects with smoking history ≥10 pack-yrs, including e-cigarettes. Former smokers with a smoking history of <10 pack-yrs must have stopped for at least 6 months prior to visit 1, including e-cigarette use.
* History of chronic alcohol or drug abuse within 12 months prior to visit 1.
* Tuberculosis requiring treatment within 12 months prior to visit 1.
* History of known immunodeficiency disorder including a positive HIV test at visit 1, or the subject is taking antiretroviral medications as determined by medical history and/or subject's verbal report.
* History of anaphylaxis or documented immune complex disease (type III hypersensitivity reactions) following any biologic therapy Subject randomized in a previous Tezepelumab study or in a current study with another investigational product.
* Pregnant, breastfeeding or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Brightling, Principal Investigator — University of Leicester, United Kingdom
Locations (28):
- United States (5):
  - Research Site, Denver, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Boston, Massachusetts
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Galveston, Texas
- Canada (6):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Hamilton, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Denmark (7):
  - Research Site, Aalborg
  - Research Site, Aarhus N
  - Research Site, Hvidovre
  - Research Site, København NV
  - Research Site, Næstved
  - Research Site, Odense C
  - Research Site, Vejle
- Germany (4):
  - Research Site, Frankfurt
  - Research Site, Frankfurt am Main
  - Research Site, Großhansdorf
  - Research Site, Landsberg
- United Kingdom (6):
  - Research Site, Cambridge
  - Research Site, Headington
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Nottingham
  - Research Site, Wythenshawe

REFERENCES:
- [Derived] Nordenmark LH, Hellqvist A, Emson C, Diver S, Porsbjerg C, Griffiths JM, Newell JD, Peterson S, Pawlikowska B, Parnes JR, Megally A, Colice G, Brightling CE. Tezepelumab and Mucus Plugs in Patients with Moderate-to-Severe Asthma. NEJM Evid. 2023 Oct;2(10):EVIDoa2300135. doi: 10.1056/EVIDoa2300135. Epub 2023 Sep 20. PMID 38320181
- [Derived] Pham TH, Chen C, Colice G, Parnes JR, Griffiths JM, Cook B. Tezepelumab normalizes serum interleukin-5 and -13 levels in patients with severe, uncontrolled asthma. Ann Allergy Asthma Immunol. 2021 Dec;127(6):689-691. doi: 10.1016/j.anai.2021.08.008. Epub 2021 Aug 14. No abstract available. PMID 34403803
- [Derived] Diver S, Khalfaoui L, Emson C, Wenzel SE, Menzies-Gow A, Wechsler ME, Johnston J, Molfino N, Parnes JR, Megally A, Colice G, Brightling CE; CASCADE study investigators. Effect of tezepelumab on airway inflammatory cells, remodelling, and hyperresponsiveness in patients with moderate-to-severe uncontrolled asthma (CASCADE): a double-blind, randomised, placebo-controlled, phase 2 trial. Lancet Respir Med. 2021 Nov;9(11):1299-1312. doi: 10.1016/S2213-2600(21)00226-5. Epub 2021 Jul 10. PMID 34256031
- [Derived] Emson C, Diver S, Chachi L, Megally A, Small C, Downie J, Parnes JR, Bowen K, Colice G, Brightling CE. CASCADE: a phase 2, randomized, double-blind, placebo-controlled, parallel-group trial to evaluate the effect of tezepelumab on airway inflammation in patients with uncontrolled asthma. Respir Res. 2020 Oct 13;21(1):265. doi: 10.1186/s12931-020-01513-x. PMID 33050900
- See also: Statistical Analysis Plan (SAP) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5180C00013&attachmentIdentifier=2a6dc7e6-ac84-4c9c-82fd-052e2347fc8f&fileName=d5180c00013-sap-ed-3-redacted.pdf&versionIdentifier=
- See also: CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5180C00013&attachmentIdentifier=e9e53dab-6b0a-4841-89a1-9e49fc805541&fileName=d5180c00013-csp-v4-redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 116 subjects randomized to Tezepelumab 210 mg Q4W or Placebo in 1:1 treatment allocation. All randomized subjects were treated.
Pre-assignment Details: The study randomized subjects across the spectrum of T2 status. Randomization was stratified by screening blood eosinophil level (<150 , 150 - <300, >=300 cells/µL).
Groups:
- Teze 210 mg Q4W: Tezepelumab subcutaneous injection
Period: Overall Study
Arm/Group | Teze 210 mg Q4W | Placebo
Started | 59 | 57
Completed | 58 | 56
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set - Include all subjects randomised to study treatment who received at least one dose of IP, irrespective of their protocol adherence and continued participation in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Teze 210 mg Q4W | Placebo | Total
Number analyzed (Participants) | 59 | 57 | 116
Age, Categorical [Count of Participants; unit: Participants] — Full Analysis Set - Include all subjects randomised to study treatment who received at least one dose of IP, irrespective of their protocol adherence and continued participation in the study.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 51 | 49 | 100
    >=65 years | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] — Full Analysis Set - Include all subjects randomised to study treatment who received at least one dose of IP, irrespective of their protocol adherence and continued participation in the study.
  Years | 50.4 (12.7) | 50.4 (13.9) | 50.4 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Full Analysis Set - Include all subjects randomised to study treatment who received at least one dose of IP, irrespective of their protocol adherence and continued participation in the study.
  Participants
    Female | 39 | 26 | 65
    Male | 20 | 31 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race - Full Analysis Set - Include all subjects randomised to study treatment who received at least one dose of IP, irrespective of their protocol adherence and continued participation in the study.
  Participants
    White | 54 | 55 | 109
    Black or African American | 2 | 1 | 3
    Asian | 2 | 1 | 3
    Other (includes Native Hawaiian or Other Pacific Islander and American Indian or Alaska Native) | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity - Full Analysis Set - Include all subjects randomised to study treatment who received at least one dose of IP, irrespective of their protocol adherence and continued participation in the study.
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 59 | 57 | 116

OUTCOME MEASURES:

1. Primary Outcome: Airway Submucosal Inflammatory Cells Ratio Change From Baseline to EOT.
Description: The change from baseline to end of treatment (EOT) expressed as a ratio i.e. (EOT/baseline) in numbers of each of the airway submucosal inflammatory cells, determined by microscopic evaluation of bronchoscopic biopsies.
Time Frame: First dose of investigational product to end of treatment (EOT) at Week 28 (or up to Week 48 due to COVID19 pandemic).
Population: Number of Participants Analyzed are all subjects randomized to study treatment who completed at least 20 weeks of study treatment and had an EOT visit not greater than 8 weeks after date of last dose of IP. In order to be included in analysis, the participants also had to have a non-missing baseline as well as a non-missing EOT assessment for the respective variable.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Teze 210 mg Q4W | Placebo
Number analyzed (Participants) | 54 | 56
Ratio
  Eosinophils: number analyzed (Participants) | 48 | 51
  Eosinophils | 0.11 [0.06 to 0.21] | 0.75 [0.41 to 1.38]
  Neutrophils: number analyzed (Participants) | 48 | 51
  Neutrophils | 1.11 [0.88 to 1.39] | 0.81 [0.66 to 1.01]
  T cells CD3+: number analyzed (Participants) | 48 | 51
  T cells CD3+ | 0.91 [0.78 to 1.07] | 0.81 [0.70 to 0.95]
  T cells CD4+: number analyzed (Participants) | 48 | 51
  T cells CD4+ | 0.96 [0.82 to 1.14] | 0.81 [0.70 to 0.95]
  Mast cells Tryptase+: number analyzed (Participants) | 48 | 51
  Mast cells Tryptase+ | 0.84 [0.70 to 1.02] | 1.01 [0.84 to 1.22]
  Mast cells Chymase+: number analyzed (Participants) | 48 | 51
  Mast cells Chymase+ | 1.07 [0.76 to 1.52] | 0.90 [0.65 to 1.26]
Statistical Analysis 1: Comparison: Teze 210 mg Q4W vs Placebo; Test type: Other; p < 0.001, ANCOVA — Nominal p-values were reported. No adjustment of multiplicity was performed; Model includes treatment+log transformed baseline value+stratification factor (screening eos count [<150, 150-<300, >=300 cells/uL]); Ratio of Geometric LSMeans = 0.15, 90% CI 2-sided [0.06 to 0.35] — Parameter : Eosinophils (cells/mm^2); 95% CI (0.05, 0.41)
Statistical Analysis 2: Comparison: Teze 210 mg Q4W vs Placebo; Test type: Other; p = 0.106, ANCOVA — Nominal p-values were reported. No adjustment of multiplicity was performed; [statistical method as in outcome 1, analysis 1]; Ratio of Geometric LSMeans = 1.36, 90% CI 2-sided [0.99 to 1.86] — Parameter: Neutrophils (cells/mm^2); 95% CI (0.94, 1.97)
Statistical Analysis 3: Comparison: Teze 210 mg Q4W vs Placebo; Test type: Other; p = 0.389, ANCOVA — Nominal p-values were reported. No adjustment of multiplicity was performed; [statistical method as in outcome 1, analysis 1]; Ratio of Geometric LSMeans = 1.12, 90% CI 2-sided [0.90 to 1.40] — Parameter: T cells CD3+ (cells/mm^2); 95% CI (0.86, 1.46)
Statistical Analysis 4: Comparison: Teze 210 mg Q4W vs Placebo; Test type: Other; p = 0.216, ANCOVA — Nominal p-values were reported. No adjustment of multiplicity was performed; [statistical method as in outcome 1, analysis 1]; Ratio of Geometric LSMeans = 1.18, 90% CI 2-sided [0.94 to 1.48] — Parameter: T cells CD4+ (cells/mm^2); 95% CI (0.90, 1.55)
Statistical Analysis 5: Comparison: Teze 210 mg Q4W vs Placebo; Test type: Other; p = 0.260, ANCOVA — Nominal p-values were reported. No adjustment of multiplicity was performed; [statistical method as in outcome 1, analysis 1]; Ratio of Geometric LSMeans = 0.83, 90% CI 2-sided [0.64 to 1.09] — Parameter: Mast cells Tryptase+ (cells/mm^2); 95% CI (0.61, 1.15)
Statistical Analysis 6: Comparison: Teze 210 mg Q4W vs Placebo; Test type: Other; p = 0.546, ANCOVA — Nominal p-values were reported. No adjustment of multiplicity was performed; [statistical method as in outcome 1, analysis 1]; Ratio of Geometric LSMeans = 1.19, 90% CI 2-sided [0.74 to 1.92] — Parameter: Mast cells Chymase+ (cells/mm^2); 95% CI (0.67, 2.10)

2. Secondary Outcome: Reticular Basement Membrane (RBM) Thickness Ratio Change From Baseline to EOT.
Description: The change from baseline to EOT expressed as a ratio i.e. (EOT/baseline) in RBM thickness, determined by microscopic evaluation of bronchoscopic biopsies.
Time Frame: First dose of investigational product to end of treatment (EOT) at Week 28 (or up to Week 48 due to COVID19 pandemic).
Population: All subjects randomised to study treatment who completed at least 20 weeks of study treatment and had a baseline assessment and an EOT assessment not greater than 8 weeks after date of last dose of IP.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Teze 210 mg Q4W | Placebo
Number analyzed (Participants) | 42 | 40
Ratio | 0.87 [0.79 to 0.95] | 0.90 [0.81 to 0.99]

3. Secondary Outcome: Percent (%) Airway Epithelial Integrity Ratio Change From Baseline to EOT.
Description: The change from baseline to EOT expressed as a ratio i.e. (EOT/baseline) in % airway epithelial, determined by microscopic evaluation of bronchoscopic biopsies.
Time Frame: First dose of investigational product to end of treatment (EOT) at Week 28 (or up to Week 48 due to COVID19 pandemic).
Population: as for outcome 1
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Teze 210 mg Q4W | Placebo
Number analyzed (Participants) | 54 | 56
Ratio
  Intact epithelium: number analyzed (Participants) | 45 | 46
  Intact epithelium | 0.87 [0.61 to 1.23] | 0.84 [0.59 to 1.19]
  Damaged epithelium: number analyzed (Participants) | 45 | 46
  Damaged epithelium | 1.01 [0.92 to 1.12] | 0.95 [0.86 to 1.04]
  Denuded epithelium: number analyzed (Participants) | 45 | 46
  Denuded epithelium | 1.05 [0.83 to 1.31] | 1.34 [1.07 to 1.68]

ADVERSE EVENTS:
Time Frame: From first dose of investigational product to end of treatment (EOT) at Week 28 (or up to Week 48 due to COVID19 pandemic).
Arm/Group | Placebo | Teze 210 mg Q4W
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/59
Serious Adverse Events (participants affected / at risk) | 7/57 | 3/59
Other Adverse Events (participants affected / at risk) | 45/57 | 48/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=57) | Teze 210 mg Q4W (N=59)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=57) | Teze 210 mg Q4W (N=59)
Dry eye (Eye disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 5 (6)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Influenza like illness (General disorders) | 3 (3) | 3 (3)
Injection site erythema (General disorders) | 2 (12) | 5 (14)
Injection site granuloma (General disorders) | 0 (0) | 2 (2)
Injection site pruritus (General disorders) | 1 (1) | 4 (5)
Oedema peripheral (General disorders) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 3 (3)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Candida infection (Infections and infestations) | 0 (0) | 2 (2)
Chronic sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Lower respiratory tract infection bacterial (Infections and infestations) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 21 (22) | 22 (28)
Oral candidiasis (Infections and infestations) | 0 (0) | 2 (4)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Rhinitis (Infections and infestations) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (5) | 3 (4)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (5)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (4)
Post procedural complication (Injury, poisoning and procedural complications) | 10 (12) | 11 (11)
Post procedural fever (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 8 (8) | 6 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 6 (9)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT03688074/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-15): https://cdn.clinicaltrials.gov/large-docs/74/NCT03688074/SAP_001.pdf